CLINICAL TRIAL: NCT02003222
Title: A Phase III Randomized Trial of Blinatumomab for Newly Diagnosed BCR-ABL-Negative B Lineage Acute Lymphoblastic Leukemia in Adults
Brief Title: Combination Chemotherapy With or Without Blinatumomab in Treating Patients With Newly Diagnosed BCR-ABL-Negative B Lineage Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02229; NCI-2013-02229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1910; PE1910_A08PAMDREVW01; E1910 (Other: ECOG-ACRIN Cancer Research Group); E1910 (Other: CTEP); U10CA021115 (NIH); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2024-09-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; B Acute Lymphoblastic Leukemia, Philadelphia Chromosome Negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Stem Cell Transplantation; Specimen Handling; blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide; Biopsy; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; Leucovorin; Spinal Puncture; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (blinatumomab, chemotherapy) (Experimental): See Detailed Description
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Biological: Blinatumomab; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Etoposide; Drug: Leucovorin Calcium; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine; Drug: Vincristine Sulfate; Procedure: X-Ray Imaging
- Arm II (chemotherapy) (Active Comparator): See Detailed Description
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Etoposide; Drug: Leucovorin Calcium; Procedure: Lumbar Puncture; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine; Drug: Vincristine Sulfate; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic SCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Blinatumomab — Given IV
  Other Names: AMG 103; AMG-103; AMG103; Anti-CD19 x Anti-CD3 Bispecific Monoclonal Antibody; Anti-CD19/Anti-CD3 Recombinant Bispecific Monoclonal Antibody MT103; Blincyto; MEDI 538; MEDI-538; MEDI538; MT 103; MT-103; MT103
  Arms: Arm I (blinatumomab, chemotherapy)
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Drug: Cytarabine — Given IT, IV, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Drug: Leucovorin Calcium — Given IV or PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given PO, IT or IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IM or IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This randomized phase III trial studies combination chemotherapy with blinatumomab to see how well it works compared to induction chemotherapy alone in treating patients with newly diagnosed breakpoint cluster region (BCR)-c-abl oncogene 1, non-receptor tyrosine kinase (ABL)-negative B lineage acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as blinatumomab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether combination chemotherapy is more effective with or without blinatumomab in treating newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the overall survival (OS) of blinatumomab in conjunction with chemotherapy to chemotherapy alone in patients with BCR-ABL-negative B cell precursor acute lymphoblastic leukemia (ALL) who are minimal residual disease (MRD) negative after induction and intensification chemotherapy, based on multiparameter flow cytometric (MFC) assessment of residual blasts.

SECONDARY OBJECTIVES:

I. To compare the relapse-free survival (RFS) of blinatumomab in conjunction with chemotherapy to chemotherapy alone in MRD negative patients after induction and intensification chemotherapy.

II. To compare the OS and RFS of those patients who are MRD positive (+) at step 3 randomization/registration and then convert to MRD negative (-) after 2 cycles of blinatumomab to those patients who are MRD- at randomization and remain MRD- after 2 cycles of blinatumomab or consolidation chemotherapy.

III. To assess the toxicities of blinatumomab in this patient population. IV. To assess the toxicities of the modified E2993 chemotherapy regimen in this patient population.

V. To describe the outcome of patients who proceed to allogeneic blood or marrow transplant after treatment with or without blinatumomab.

LABORATORY OBJECTIVES:

I. To determine differences in MRD kinetics among patients with the BCR/ABL1-like B-lineage ALL, and to compare the OS (and RFS) of patients with BCR-ABL-like phenotype with those without BCR-ABL-like phenotype.

II. To evaluate the incidence of anti-blinatumomab antibody formation.

OUTLINE:

INDUCTION CHEMOTHERAPY: Patients receive cytarabine intrathecally (IT) on day 1; daunorubicin hydrochloride intravenously (IV) over 10-15 minutes on days 1, 8, 15, and 22; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone orally (PO) daily on days 1-7 (and 15-21 for patients age < 55 years only); methotrexate IT on day 14; pegaspargase intramuscularly (IM) or IV on day 18 (patients age < 55 years); and CD20 positive patients may optionally receive rituximab IV on day 8 and 15. Beginning on day 29, patients with absolute neutrophil count (ANC) >= 0.75 x 10^9/L and platelets > 75 x 10^9/L (patients with delayed hematologic recovery) (patients with residual disease that is delaying count begin treatment immediately) receive cyclophosphamide IV over 30 minutes on days 1 and 29, cytarabine IV over 30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14, 29-42, pegaspargase IM or IV on day 15 (patients age < 55 years), patients receiving treatment for central nervous system (CNS) 2 or 3 leukemia in cycle 1 receive methotrexate IT on days 1, 8, 15, and 22, and CD20 positive patients may optionally receive rituximab IV on days 8 and 15.

INTENSIFICATION THERAPY: Beginning 4 weeks after the completion of cycle 2 of induction therapy, patients receive intensification therapy comprising high-dose methotrexate IV over 2 hours on days 1 and 8, and pegaspargase IM or IV on day 9.

Patients are then randomized to 1 of 2 treatment arms.

Patients randomized to the blinatumomab group receive blinatumomab IV continuously on days 1-28. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may then undergo allogeneic stem cell transplant (SCT) or proceed to consolidation therapy per investigator discretion.

CONSOLIDATION THERAPY: Beginning after the second cycle of blinatumomab (patients randomized to the blinatumomab group) or after intensification therapy (patients not randomized to blinatumomab), patients receive cytarabine IV over 30 minutes or SC on days 1-5, etoposide IV over 1 hour on days 1-5, methotrexate IT on day 1, and pegaspargase IM or IV on day 5, and CD20 positive patients may optionally receive rituximab IV on day 5. Beginning 4 weeks from day 1 of cycle 1, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may receive rituximab as in cycle 1. Beginning 4 weeks from day 1 of cycle 2, patients receive daunorubicin hydrochloride IV over 10-15 minutes on day 1, 8, 15, and 22; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone PO daily on days 1-7 (and 15-21 for patients age < 55 years); methotrexate IT on day 2; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 30 minutes or SC on days 30-33 and 37-40; mercaptopurine PO on days 29-42 and CD20 positive patients may receive rituximab on day 8. Beginning 8 weeks from day 1 of cycle 3, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may optionally receive rituximab as in cycle 1. Patients randomized to blinatumomab repeat cycle 4 and then receive blinatumomab IV continuously on days 1-28.

MAINTENANCE THERAPY: Within 6 weeks after beginning last cycle of consolidation therapy, patients receive mercaptopurine PO daily, methotrexate PO or IV over 2 hours once weekly for 2.5 years, vincristine sulfate IV on day 1 every 3 months, prednisone PO on days 1-5 every 3 months, and methotrexate IT on day 1 every 3 months. Treatment continues for up to 2.5 years in the absence of disease progression or unacceptable toxicity.

Patients undergo x-ray imaging during screening, lumbar puncture while on study, and bone marrow aspiration, bone marrow biopsy, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then every 12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION
* Diagnostic bone marrow and/or peripheral blood specimens must be submitted for immunophenotyping and selected molecular testing, and the establishment of BCR/ABL status; testing will be performed by the Eastern Cooperative Oncology Group (ECOG)-American College of Radiation Imaging Network (ACRIN) Leukemia Translational Research Laboratory (LTRL) and reported to the institution

  * NOTE: IT IS ESSENTIAL THAT A SAMPLE CONTAINING SUFFICIENT BLAST CELLS BE SUBMITTED TO THE ECOG-ACRIN LTRL AT BASELINE SO THAT SUBSEQUENT BONE MARROW ASSESSMENTS OF MRD CAN BE DONE; IN ADDITION TO ALLOWING THE LTRL TO CONFIRM ELIGIBILITY BASED ON BLAST CELL IMMUNOPHENOTYPE AND BCR/ABL STATUS, IT IS ALSO IMPERATIVE THAT AN ADEQUATE NUMBER OF BLASTS BE BANKED FOR ANALYSIS BY DRS MULLIGHAN/WILLMAN. WITHOUT ADEQUATE BASELINE SAMPLES, PATIENTS WILL NOT BE ABLE TO BE TREATED AND RANDOMIZED ON THIS PROTOCOL; IF A BONE MARROW ASPIRATE IS NOT AVAILABLE FOR LTRL SUBMISSION AT BASELINE, IT IS IMPERATIVE THAT DR PAIETTA FROM THE LTRL IS CALLED TO DISCUSS THE PERIPHERAL BLOOD WHITE BLOOD CELL (WBC) AND BLAST COUNT BEFORE BLOOD ONLY IS SUBMITTED
  * NOTE: Hydroxyurea can be given for up to 5 days prior to initiation of protocol therapy for control of leukocyte count and/or other symptoms or signs; corticosteroids can be given after pre-registration to the protocol and submission of baseline marrow and blood samples for control of leukocyte count and/or other symptoms or signs prior to initiation of protocol therapy if needed; if corticosteroids are given prior to pre-registration, contact the study chair as the patient may still be eligible to participate
* INDUCTION ELIGIBILITY CRITERIA-STEP 1
* Age >= 30 years and =< 70 years
* New diagnosis of B lineage ALL must be made upon bone marrow or peripheral blood immunophenotyping; cases with myeloid antigen expression, but unequivocal lymphoid immunophenotype, are eligible
* Negativity for the Philadelphia chromosome must be established by conventional cytogenetics, fluorescence in situ hybridization (FISH) and/or polymerase chain reaction (PCR); patients who are negative for the Philadelphia chromosome by conventional cytogenetics must have FISH or PCR performed for BCR/ABL to exclude occult translocations
* Cytogenetic analysis must be performed from diagnostic bone marrow (preferred) or if adequate number of circulating blasts from peripheral blood; FISH testing for common B-lineage ALL abnormalities including t(9;22) (BCR/ABL1), t(12;21) (ETS-variant gene 6 [ETV6]/runt-related transcription factor 1 [RUNX1]), t(1;19) (pre-B-cell leukemia homeobox 1 [PBX1]/transcription factor 3 [TCF3]), +4,+10,+17, (centromeric [Cen]4/Cen10/Cen17), t(11q23;var), (myeloid/lymphoid or mixed lineage leukemia [MLL]), deletion (del)(9p) (cyclin-dependent kinase inhibitor 2A [CDKN2A]/Cen9), and t(14;var) (immunoglobulin heavy chain [IGH] is encouraged); if there are few or no circulating blasts and an adequate marrow sample cannot be obtained for cytogenetic analysis, the patient may still enroll on the trial
* Serum direct bilirubin < 2 mg/dl or serum total bilirubin =< 3 (obtained =< 48 hours prior to registration); NOTE: the above stipulation for normal hepatic function does not apply if liver dysfunction is due to leukemia infiltration
* Serum creatinine < 2 mg/dl (obtained =< 48 hours prior to registration); NOTE: the above stipulation for normal hepatic function does not apply if liver dysfunction is due to leukemia infiltration
* Patient should be human leukocyte antigen (HLA) typed (A, B, C, DR and DQ) during induction therapy phase or a written explanation for not undergoing HLA typing on the flow sheet
* Patients with known human immunodeficiency virus (HIV) infection are eligible if they meet all of the following criteria:

  * No history of acquired immune deficiency syndrome (AIDS)-related complications other than a history of low CD4+ T-cell count (< 200/mm^3) prior to initiation of combination antiretroviral therapy; on study CD4+ T-cell count may not be informative due to leukemia and should not be used as an exclusion criterion if low
  * Patient must be healthy on the basis of HIV disease with high likelihood of near normal life span were it not for the leukemia
  * Patient must have serum HIV viral load of < 200 copies/mm^3
  * Patient must be on combination antiretroviral therapy with minimal pharmacokinetic interactions with study therapy and minimal overlapping clinical toxicity with protocol therapy
  * Patient must not be receiving protease inhibitors or once daily formulations containing cobicistat, stavudine, or on regimens containing stavudine or zidovudine
  * It is recommended to utilize a regimen of the integrase inhibitor, dolutegravir, combined with either disoproxil fumarate/emtricitabine or dolutegravir combined with tenofovir alafenamide/emtricitabine
* Patient must have no history of recent myocardial infarction (within three months), uncontrolled congestive heart failure, or uncontrolled cardiac arrhythmia
* Patient must have a normal cardiac ejection fraction by pretreatment multigated acquisition scan (MUGA) or echocardiogram within 4 weeks prior to registration (resting ejection fraction >= 40% or >= 5% increase with exercise), shortening fraction by echocardiogram >= 24%, or to within the normal range of values for the institution
* Women must not be pregnant or breast-feeding due to administration of teratogenic chemotherapy and must not become pregnant or breastfeed during protocol therapy and for at least 3 months after protocol therapy; woman of childbearing potential must abstain from sexual activity or be willing to use 2 highly effective forms of contraception throughout protocol therapy and for at least an additional 3 months after the last dose of protocol-specified therapy; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Men who have a female partner of childbearing potential must be willing to use 2 highly effective forms of contraception throughout protocol therapy and for at least an additional 3 months after the last dose of protocol-specified therapy; men who have a pregnant partner must be willing to use a condom during sexual activity throughout protocol therapy and for 3 months after the last dose of protocol-specified therapy
* ECOG performance score 0-3
* Patient must have given written informed consent
* POST-INDUCTION THERAPY ELIGIBILITY CRITERIA (PRIOR TO INTENSIFICATION-STEP 2)
* ECOG performance status 0-2
* Patients must have achieved a CR or CRi
* Patients who have achieved a CR or CRi must have maintained peripheral blood evidence of a CR or CRi
* Patient must be CNS (cerebrospinal fluid [CSF]) negative for leukemia
* Patients must have resolved any serious infectious complications related to induction
* Any significant medical complications related to induction must have resolved
* Serum creatinine =< 2.0 mg/dl (obtained =< 48 hours prior to registration)
* Serum direct bilirubin < 2 mg/dL or serum total bilirubin =< 3 (obtained =< 48 hours prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x upper limit of normal (ULN) (obtained =< 48 hours prior to registration)
* RANDOMIZATION OR ASSIGNMENT TO BLINATUMOMAB OR NO BLINATUMOMAB-STEP 3
* Patients must have an ECOG performance status of 0-2
* Patients must have maintained peripheral blood evidence of a remission and must have a CR or CRi, confirmed on restaging bone marrow (BM) aspirate and biopsy
* Patients must have resolved any serious infectious complications related to therapy
* Any significant medical complications related to therapy must have resolved
* Direct or total bilirubin < 1.5 x ULN (unless related to Gilbert's or Meulengracht's syndrome); the values must be obtained within 48 hours prior to randomization
* Serum creatinine < 1.5 x ULN; the values must be obtained within 48 hours prior to randomization
* Bone marrow aspirates must be submitted for centralized minimal residual disease (MRD) assessment performed by the ECOG-ACRIN Leukemia Translational Research Laboratory
* MRD results will be reported to the submitting institution

  * NOTE: FOR MRD ASSESSMENTS, AN ASPIRATE FROM A SEPARATE BONE MARROW ASPIRATION SITE MUST BE SUBMITTED (THE NEEDLE CAN BE RE-DIRECTED THROUGH THE SAME SKIN PUNCTURE SITE); ONLY SUBMIT ASPIRATES FROM THE FIRST PULL OF AN ASPIRATION SITE FOR MRD TESTING; DO NOT SUBMIT SAMPLES FROM THE SECOND OR THIRD PULL OF THE SAME ASPIRATION SITE
  * In B-lineage ALL, MRD levels in peripheral blood or from a dilute marrow aspiration can be 300% lower, on average, than those in bone marrow at a given time point; submitting a first pull from a separate aspiration site will ensure that MRD determinations used in randomization and trial interpretation are accurate

    * NOTE: failure to submit bone marrow aspirates will result in a major violation at the time of an audit
* CRITERIA FOR ALLOGENEIC TRANSPLANTATION
* A suitable donor must be identified; there are no restrictions on donor type and can include a matched sibling, a matched or mismatched unrelated donor, a family haplotype matched donor or a cord blood donor (single or double)
* Patients should meet the eligibility criteria for RANDOMIZATION OR ASSIGNMENT TO BLINATUMOMAB OR NO BLINATUMOMAB-STEP 3
* Patients must be considered reliable enough to comply with the medication regimen and follow-up, and have social support necessary to allow this compliance
* CRITERIA FOR MAINTENANCE THERAPY-STEP 4: Patients must have an ECOG performance status of 0-3
* CRITERIA FOR MAINTENANCE THERAPY-STEP 4: Patients must have maintained peripheral blood evidence of a remission and must have a CR or CRi, confirmed on restaging BM aspirate and biopsy
* CRITERIA FOR MAINTENANCE THERAPY-STEP 4: Patients must have resolved any serious infectious complications related to therapy
* CRITERIA FOR MAINTENANCE THERAPY-STEP 4: Any significant medical complications related to therapy must have resolved

Exclusion Criteria:

* Mature B ALL (Burkitt's-like leukemia) is excluded from enrollment in this trial; pre-study bone marrow biopsy and aspirate must be completed =< 1 week prior to registration
* Patient must not have a concurrent active malignancy for which they are receiving treatment
* Patient must not have intercurrent organ damage or medical problems that will jeopardize the outcome of therapy (i.e., psychiatric disorder, drug abuse, pregnancy)
* Patient must not have an antecedent hematologic disorder
* Patient must not have a history or presence of clinically relevant central nervous system (CNS) pathology such as epilepsy, seizure, paresis, aphasia, stroke, severe brain injuries, dementia; Parkinson's disease, cerebellar disease, organic brain syndrome, psychosis, or other significant CNS abnormalities
* Patient must not have an active uncontrolled infection

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Litzow, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (546):
- United States (533):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner High Grove, Baton Rouge, Louisiana
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (6):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Clinical Research Unit at Vancouver Coastal Health Authority, Vancouver, British Columbia
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Litzow MR, Sun Z, Mattison RJ, Paietta EM, Roberts KG, Zhang Y, Racevskis J, Lazarus HM, Rowe JM, Arber DA, Wieduwilt MJ, Liedtke M, Bergeron J, Wood BL, Zhao Y, Wu G, Chang TC, Zhang W, Pratz KW, Dinner SN, Frey N, Gore SD, Bhatnagar B, Atallah EL, Uy GL, Jeyakumar D, Lin TL, Willman CL, DeAngelo DJ, Patel SB, Elliott MA, Advani AS, Tzachanis D, Vachhani P, Bhave RR, Sharon E, Little RF, Erba HP, Stone RM, Luger SM, Mullighan CG, Tallman MS. Blinatumomab for MRD-Negative Acute Lymphoblastic Leukemia in Adults. N Engl J Med. 2024 Jul 25;391(4):320-333. doi: 10.1056/NEJMoa2312948. PMID 39047240
- [Derived] Seftel MD. Hyper-CVAD: a regimen for all seasons. Lancet Haematol. 2020 Jul;7(7):e501-e502. doi: 10.1016/S2352-3026(20)30179-4. No abstract available. PMID 32589970

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 17, 2013 and closed to accrual on October 15, 2019 after enrolling a total of 488 patients.
Groups:
- MRD Negative - Blinatumomab + Chemotherapy: MRD negative patients received induction treatment and intensification treatment and then were randomized to receive blinatumomab plus chemotherapy.
- MRD Negative - Chemotherapy: MRD negative patients received induction treatment and intensification treatment and then were randomized to receive chemotherapy.
- MRD Positive - Blinatumomab + Chemotherapy: MRD positive patients received induction treatment and intensification treatment and then were randomized or assigned to receive blinatumomab plus chemotherapy.
- MRD Positive - Chemotherapy: MRD positive patients received induction treatment and intensification treatment and then were randomized to receive chemotherapy.
- No Randomization/Registration: Patients were registered to receive induction treatment and intensification treatment but did not enter the randomization part of the study.
Period: Induction
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy | MRD Positive - Blinatumomab + Chemotherapy | MRD Positive - Chemotherapy | No Randomization/Registration
Started | 112 | 112 | 40 | 22 | 202
Received Treatment and Adverse Event Assessment Available | 112 | 112 | 40 | 22 | 193
Completed | 112 | 112 | 40 | 22 | 47
Not Completed | 0 | 0 | 0 | 0 | 155
Not completed — Never started treatment | 0 | 0 | 0 | 0 | 8
Not completed — Complete remission or complete remission incomplete not achieved | 0 | 0 | 0 | 0 | 67
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 13
Not completed — Alternative therapy | 0 | 0 | 0 | 0 | 12
Not completed — Disease progression | 0 | 0 | 0 | 0 | 22
Not completed — Death | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 8
Not completed — Other reasons | 0 | 0 | 0 | 0 | 22
Period: Intensification
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy | MRD Positive - Blinatumomab + Chemotherapy | MRD Positive - Chemotherapy | No Randomization/Registration
Started | 112 | 112 | 40 | 22 | 47
Received Treatment and Adverse Event Assessment Available | 112 | 112 | 40 | 22 | 30
Completed | 112 | 112 | 40 | 22 | 0
Not Completed | 0 | 0 | 0 | 0 | 47
Not completed — Never started treatment | 0 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 6
Not completed — Alternative therapy | 0 | 0 | 0 | 0 | 8
Not completed — Disease progression | 0 | 0 | 0 | 0 | 18
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5
Not completed — Other reasons | 0 | 0 | 0 | 0 | 8
Period: Randomization/Registration
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy | MRD Positive - Blinatumomab + Chemotherapy | MRD Positive - Chemotherapy | No Randomization/Registration
Started | 112 | 112 | 40 | 22 | 0
Received Treatment and Adverse Event Assessment Available | 111 | 110 | 35 | 16 | 0
Completed | 112 | 112 | 40 | 22 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Maintenance
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy | MRD Positive - Blinatumomab + Chemotherapy | MRD Positive - Chemotherapy | No Randomization/Registration
Started | 67 | 69 | 13 | 2 | 0
Received Treatment and Adverse Event Assessment Available | 66 | 68 | 12 | 2 | 0
Completed | 67 | 69 | 13 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy | MRD Positive - Blinatumomab + Chemotherapy | MRD Positive - Chemotherapy | No Randomization/Registration | Total
Number analyzed (Participants) | 112 | 112 | 40 | 22 | 202 | 488
Age, Continuous [Median (Full Range); unit: years] | 51.5 [30 to 69] | 50 [30 to 70] | 49 [30 to 68] | 54.5 [30 to 69] | 52 [30 to 70] | 51 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 26 | 8 | 90 | 237
  Male | 55 | 56 | 14 | 14 | 112 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 8 | 5 | 34 | 70
  Not Hispanic or Latino | 95 | 95 | 30 | 16 | 155 | 391
  Unknown or Not Reported | 4 | 7 | 2 | 1 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 5 | 8
  Asian | 3 | 2 | 1 | 0 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 9 | 4 | 3 | 1 | 6 | 23
  White | 87 | 89 | 30 | 21 | 164 | 391
  More than one race | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 10 | 16 | 6 | 0 | 21 | 53

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Among Patients Who Were MRD Negative After Induction and Intensification Chemotherapy
Description: Overall survival is defined as the time from randomization to death of any cause.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: All MRD-negative patients randomized to either blinatumomab + chemotherapy or chemotherapy alone were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy
Number analyzed (Participants) | 112 | 112
months | NA [NA to NA] — Median OS not reached The 95% confidence intervals were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [66.5 to NA] — Median OS not reached The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: MRD Negative - Blinatumomab + Chemotherapy vs MRD Negative - Chemotherapy; Test type: Superiority; p = 0.003, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.25 to 0.76] — hazard ratio: blinatumomab + chemotherapy vs. chemotherapy alone

2. Secondary Outcome: Relapse-free Survival (RFS) Among Patients Who Were MRD Negative After Induction and Intensification Chemotherapy
Description: RFS was defined as time from randomization to relapse or to death without documentation of relapse. Patients without events were censored at the date of last disease assessment.
  Relapse/Persistent Disease
  Persistent disease/Relapse following complete remission (CR)/complete remission incomplete (CRi) is defined as:
  * Reappearance or persistence of blasts in the blood
  * Presence of > 5% blasts, not attributable to another cause (e.g., bone marrow regeneration).
  * In the case of isolated CNS relapse such as a positive cytospin examination of CSF, please consult with Study Chair. Perform bone marrow biopsy (if not already done) to confirm presence or lack of medullary relapse.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MRD Negative - Blinatumomab + Chemotherapy | MRD Negative - Chemotherapy
Number analyzed (Participants) | 112 | 112
months | NA [37.1 to NA] — Median RFS not reached The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 35.2 [30.3 to 69.0]
Statistical Analysis 1: Comparison: MRD Negative - Blinatumomab + Chemotherapy vs MRD Negative - Chemotherapy; Test type: Superiority; p = 0.015, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.31 to 0.89] — hazard ratio: Blinatumomab + Chemotherapy vs. Chemotherapy alone

3. Secondary Outcome: RFS Among of Those Who Are MRD+ at Randomization and Then Convert to MRD- After 2 Cycles of Blinatumomab to Those Patients Who Are MRD- at Randomization and Remain MRD- After 2 Cycles of Blinatumomab or Consolidation Chemotherapy
Description: RFS was defined as time from end of 2 cycles of blinatumomab to relapse or to death without documentation of relapse. Patients without events were censored at the date of last disease assessment.
  Relapse/Persistent Disease
  Persistent disease/Relapse following complete remission (CR)/complete remission incomplete (CRi) is defined as:
  * Reappearance or persistence of blasts in the blood
  * Presence of > 5% blasts, not attributable to another cause (e.g., bone marrow regeneration).
  * In the case of isolated CNS relapse such as a positive cytospin examination of CSF, please consult with Study Chair. Perform bone marrow biopsy (if not already done) to confirm presence or lack of medullary relapse.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: Patients with MRD data at the end of 2 cycles of blinatumomab were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MRD+ Then Convert to MRD-: Patients who are MRD positive (MRD+) at randomization/registration and then convert to MRD negative (MRD-) after 2 cycles of blinatumomab or consolidation chemotherapy.
  .
- MRD- Then Remain MRD-: Patients who are MRD negative (MRD-) at randomization/registration and then remain MRD negative (MRD-) after 2 cycles of blinatumomab or consolidation chemotherapy.
  .
Arm/Group | MRD+ Then Convert to MRD- | MRD- Then Remain MRD-
Number analyzed (Participants) | 28 | 89
months | NA [NA to NA] — Median RFS not reached The 95% confidence intervals were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [38.9 to NA] — Median RFS not reached The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: MRD+ Then Convert to MRD- vs MRD- Then Remain MRD-; Test type: Superiority; p = 0.67, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.22 to 2.65]

4. Secondary Outcome: OS Among of Those Who Are MRD+ at Randomization and Then Convert to MRD- After 2 Cycles of Blinatumomab to Those Patients Who Are MRD- at Randomization and Remain MRD- After 2 Cycles of Blinatumomab or Consolidation Chemotherapy
Description: OS was defined as time from end of 2 cycles of blinatumomab to death of any cause
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: Patients with MRD data at the end of 2 cycles of blinatumomab were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MRD+ Then Convert to MRD- | MRD- Then Remain MRD-
Number analyzed (Participants) | 28 | 89
months | NA [NA to NA] — Median OS not reached The 95% confidence intervals were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — Median OS not reached The 95% confidence intervals were not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: MRD+ Then Convert to MRD- vs MRD- Then Remain MRD-; Test type: Superiority; p = 1.00, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.28 to 3.63]

5. Secondary Outcome: OS Among MRD Negative Patients Who Proceed to Allogeneic Transplant on Study
Description: OS was defined as time from allogeneic transplant to death of any cause.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Population: MRD negative patients who proceeded to allogeneic transplant after treatment with blinatumomab plus chemotherapy or chemotherapy alone were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- MRD Negative Patients Receiving Blinatumomab + Chemotherapy and Then Allogeneic Transplant: Patients who proceed to allogeneic blood or marrow transplant after treatment with blinatumomab and chemotherapy.
- MRD Negative Patients Receiving Chemotherapy and Then Allogeneic Transplant: Patients who proceed to allogeneic blood or marrow transplant after treatment with chemotherapy.
  .
Arm/Group | MRD Negative Patients Receiving Blinatumomab + Chemotherapy and Then Allogeneic Transplant | MRD Negative Patients Receiving Chemotherapy and Then Allogeneic Transplant
Number analyzed (Participants) | 22 | 22
months | NA [NA to NA] — Median OS not reached The 95% confidence intervals were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [30.2 to NA] — Median OS not reached The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: MRD Negative Patients Receiving Blinatumomab + Chemotherapy and Then Allogeneic Transplant vs MRD Negative Patients Receiving Chemotherapy and Then Allogeneic Transplant; Test type: Superiority; p = 0.41, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.17 to 2.11] — hazard ratio: blinatumomab + chemotherapy vs. chemotherapy alone

6. Other Pre Specified Outcome: To Determine Differences in MRD Kinetics Among Patients With the BCR/ABL1-like B-lineage ALL, and to Compare the OS (and RFS) of Patients With BCR-ABL-like Phenotype With Those Without BCR-ABLlike Phenotype
Description: To determine differences in MRD kinetics among patients with the BCR/ABL1-like B-lineage ALL, and to compare the OS (and RFS) of patients with BCR-ABL-like phenotype with those without BCR-ABLlike phenotype
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 3 years, then annually for 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Incidence of Anti-blinatumomab Antibody Formation
Description: To evaluate the incidence of anti-blinatumomab antibody formation
Time Frame: Assessed at baseline, end of 2 cycles of blinatumomab, end of 4 cycles of blinatumomab, and end of blinatumomab treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every while on treatment and for 30 days after the end of treatment, up to 9 years
Description: Patients who received treatment and were assessed for adverse events are included in the analysis of serious adverse events as well as other adverse events.
Groups:
- Induction: Patients receive cytarabine intrathecally (IT) on day 1; daunorubicin hydrochloride intravenously (IV) over 10-15 minutes on days 1, 8, 15, and 22; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone orally (PO) daily on days 1-7 (and 15-21 for patients age < 55 years only); methotrexate IT on day 14; pegaspargase intramuscularly (IM) or IV on day 18 (patients age < 55 years); and CD20 positive patients may optionally receive rituximab IV on day 8 and 15. Beginning on day 29, patients with absolute neutrophil count (ANC) >= 0.75 x 10^9/L and platelets > 75 x 10^9/L (patients with delayed hematologic recovery) (patients with residual disease that is delaying count begin treatment immediately) receive cyclophosphamide IV over 30 minutes on days 1 and 29, cytarabine IV over 30 minutes or subcutaneously (SC) on days 1-4, 8-11, 29-32, and 36-39, mercaptopurine PO on days 1-14, 29-42, pegaspargase IM or IV on day 15 (patients age < 55 years), patients receiving treatment for central nervous system (CNS) 2 or 3 leukemia in cycle 1 receive methotrexate IT on days 1, 8, 15, and 22, and CD20 positive patients may optionally receive rituximab IV on days 8 and 15.
- Intensification: Beginning 4 weeks after the completion of cycle 2 of induction therapy, patients receive intensification therapy comprising high-dose methotrexate IV over 2 hours on days 1 and 8, and pegaspargase IM or IV on day 9.
- Blinatumomab: Patients receive blinatumomab IV continuously on days 1-28. Treatment repeats every 6 weeks for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients may then undergo allogeneic stem cell transplant (SCT) or proceed to consolidation therapy per investigator discretion.
  Consolidation therapy: Beginning after the second cycle of blinatumomab, patients receive cytarabine IV over 30 minutes or SC on days 1-5, etoposide IV over 1 hour on days 1-5, methotrexate IT on day 1, and pegaspargase IM or IV on day 5, and CD20 positive patients may optionally receive rituximab IV on day 5. Beginning 4 weeks from day 1 of cycle 1, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may receive rituximab as in cycle 1. Beginning 4 weeks from day 1 of cycle 2, patients receive daunorubicin hydrochloride IV over 10-15 minutes on day 1, 8, 15, 22; vincristine sulfate IV on days 1, 8, 15, 22; dexamethasone PO daily on days 1-7 (and 15-21 for patients age < 55 years); methotrexate IT on day 2; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 30 minutes or SC on days 30-33 and 37-40; mercaptopurine PO on days 29-42 and CD20 positive patients may receive rituximab on day 8. Beginning 8 weeks from day 1 of cycle 3, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may optionally receive rituximab as in cycle 1. Patients repeat cycle 4 and then receive blinatumomab IV continuously on days 1-28.
- No Blinatumomab: Patients undergo allogeneic stem cell transplant (SCT) or proceed to consolidation therapy per investigator discretion.
  Consolidation therapy: After intensification therapy, patients receive cytarabine IV over 30 minutes or SC on days 1-5, etoposide IV over 1 hour on days 1-5, methotrexate IT on day 1, and pegaspargase IM or IV on day 5, and CD20 positive patients may optionally receive rituximab IV on day 5. Beginning 4 weeks from day 1 of cycle 1, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may receive rituximab as in cycle 1. Beginning 4 weeks from day 1 of cycle 2, patients receive daunorubicin hydrochloride IV over 10-15 minutes on day 1, 8, 15, and 22; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone PO daily on days 1-7 (and 15-21 for patients age < 55 years); methotrexate IT on day 2; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV over 30 minutes or SC on days 30-33 and 37-40; mercaptopurine PO on days 29-42 and CD20 positive patients may receive rituximab on day 8. Beginning 8 weeks from day 1 of cycle 3, patients receive cytarabine, etoposide, methotrexate, and CD20 positive patients may optionally receive rituximab as in cycle 1.
- Maintenance: Within 6 weeks after beginning last cycle of consolidation therapy, patients receive mercaptopurine PO daily, methotrexate PO or IV over 2 hours once weekly for 2.5 years, vincristine sulfate IV on day 1 every 3 months, prednisone PO on days 1-5 every 3 months, and methotrexate IT on day 1 every 3 months. Treatment continues for up to 2.5 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Induction | Intensification | Blinatumomab | No Blinatumomab | Maintenance
All-Cause Mortality (participants affected / at risk) | 103/479 | 28/316 | 23/146 | 31/126 | 27/148
Serious Adverse Events (participants affected / at risk) | 457/479 | 166/316 | 134/146 | 121/126 | 121/148
Other Adverse Events (participants affected / at risk) | 227/479 | 153/316 | 94/146 | 65/126 | 93/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (N=479) | Intensification (N=316) | Blinatumomab (N=146) | No Blinatumomab (N=126) | Maintenance (N=148)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 244 | 56 | 38 | 50 | 17
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 124 | 1 | 31 | 34 | 10
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 5 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 2 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0
Edema limbs (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 29 | 4 | 5 | 5 | 3
Fever (General disorders) | 6 | 0 | 2 | 1 | 0
Flu like symptoms (General disorders) | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (General disorders) | 5 | 0 | 1 | 0 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 4 | 3 | 2 | 2
Anal mucositis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 3 | 5 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 5 | 2 | 1 | 4 | 5
Nausea (Gastrointestinal disorders) | 19 | 4 | 6 | 2 | 3
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 9 | 4 | 0 | 1 | 3
Proctitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Rectal mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Small intestinal mucositis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Typhlitis (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 17 | 0 | 3 | 4 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 4 | 1 | 0 | 1 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 2 | 0 | 0 | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 1 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 6 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 0 | 0 | 0 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bone infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 9 | 3 | 4 | 5 | 0
Endocarditis infective (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 4 | 0 | 2 | 0 | 0
Esophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 17 | 1 | 3 | 2 | 4
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pancreas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 22 | 2 | 8 | 9 | 1
Sinusitis (Infections and infestations) | 4 | 0 | 2 | 1 | 0
Skin infection (Infections and infestations) | 5 | 1 | 1 | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 1 | 4 | 1
Urinary tract infection (Infections and infestations) | 10 | 0 | 2 | 1 | 4
Infections and infestations - Other, specify (Infections and infestations) | 14 | 0 | 5 | 4 | 6
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 56 | 15 | 8 | 7 | 29
Alkaline phosphatase increased (Investigations) | 16 | 3 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 30 | 9 | 5 | 3 | 10
Blood bilirubin increased (Investigations) | 52 | 6 | 2 | 2 | 11
Cholesterol high (Investigations) | 1 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1
Fibrinogen decreased (Investigations) | 18 | 2 | 1 | 1 | 0
GGT increased (Investigations) | 7 | 1 | 3 | 1 | 0
Lipase increased (Investigations) | 5 | 4 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 133 | 37 | 39 | 35 | 23
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 423 | 85 | 118 | 116 | 88
Platelet count decreased (Investigations) | 385 | 35 | 93 | 95 | 36
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 2 | 0 | 0
Weight loss (Investigations) | 1 | 1 | 0 | 1 | 0
White blood cell decreased (Investigations) | 397 | 23 | 65 | 78 | 49
Investigations - Other, specify (Investigations) | 0 | 1 | 1 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 0 | 2 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 1 | 3 | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 38 | 16 | 9 | 9 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 19 | 7 | 4 | 5 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 20 | 1 | 2 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 1 | 2 | 3 | 0
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 23 | 2 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Arachnoiditis (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 7 | 0 | 0
Encephalopathy (Nervous system disorders) | 5 | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 24 | 2 | 6 | 6 | 2
Intracranial hemorrhage (Nervous system disorders) | 2 | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 2 | 4
Seizure (Nervous system disorders) | 2 | 0 | 2 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 4 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 4 | 0 | 4 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 5 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 0 | 4 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 4 | 0 | 6 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 0 | 3 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 17 | 4 | 3 | 1 | 2
Hypotension (Vascular disorders) | 13 | 1 | 3 | 0 | 0
Thromboembolic event (Vascular disorders) | 22 | 2 | 2 | 3 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (N=479) | Intensification (N=316) | Blinatumomab (N=146) | No Blinatumomab (N=126) | Maintenance (N=148)
Anemia (Blood and lymphatic system disorders) | 42 | 83 | 67 | 38 | 60
Fatigue (General disorders) | 35 | 0 | 16 | 7 | 18
Fever (General disorders) | 0 | 0 | 14 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 37 | 18 | 7 | 11 | 15
Constipation (Gastrointestinal disorders) | 34 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 72 | 24 | 28 | 19 | 20
Nausea (Gastrointestinal disorders) | 44 | 19 | 16 | 6 | 13
Vomiting (Gastrointestinal disorders) | 100 | 32 | 32 | 22 | 13
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 16 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 8 | 3 | 19
Aspartate aminotransferase increased (Investigations) | 26 | 16 | 0 | 0 | 16
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 10
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 14
Neutrophil count decreased (Investigations) | 0 | 42 | 33 | 4 | 40
Platelet count decreased (Investigations) | 39 | 70 | 56 | 27 | 55
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 14
Headache (Nervous system disorders) | 124 | 27 | 44 | 26 | 23
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 9 | 3 | 17
Tremor (Nervous system disorders) | 0 | 0 | 19 | 2 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 8 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02003222/Prot_SAP_000.pdf